CLINICAL TRIAL: NCT06552533
Title: Comparison of Resistance Training With and Without Plyometric Exercises on Pain, Range of Motion, Dynamic Balance and Strength Among Athletes With Chronic Ankle Instability.
Brief Title: Comparison of Resistance Training With and Without Plyometric Exercises on Athletes With Chronic Ankle Instability.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0473
Record Dates: First submitted 2024-06-24; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Chronic Ankle Instability
Keywords: goniometry, plyometric exercises, resistance training
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: the investigator and participant will be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Exercises with Plyometric exercises (Experimental): We will apply protocol for 8 weeks 24 Sessions (3 sessions in a week). Resistive training will start in the form of manual resistive exercise for dorsiflexion, plantar flexion, eversion and inversion (manual resistance was applied for 3 to 5 seconds for ten repetitions in each cardinal plane). While controlling the time that a maximal contraction will maintained, the therapist will assure that the targeted musculature will being maximally loaded. Resistance will be applied to the dorsum of the foot just above the toes to resist dorsiflexion and to the plantar surface of the foot at the metatarsals to resist plantar flexion. After resistance training the athletes will go for plyometric exercises and will follow the following guidelines.Tubing Exercises and Plyometric Ankle Jumps Ankle Circles. Move just your foot and ankle, not your leg. Vary the stretch by tracing out the letters of the alphabet with your big toe.
  Interventions: Other: Resistance Exercises with Plyometric exercises
- Resistance Exercises without Plyometric exercises (Active Comparator): We will apply protocol for 8 weeks 24 Sessions (3 sessions in a week).We will apply protocol for 8 weeks 24 Sessions (3 sessions in a week) and 10 sec rest between each segment, 3 sets of 10 repetitions. Resistive training will start in the form of manual resistive exercise for dorsiflexion, plantar flexion, eversion and inversion (manual resistance was applied for 3 to 5 seconds for ten repetitions in each cardinal plane). Active weight bearing exercises in the form of heel rise and toe rise will performed for ten repetitions each. Towel curl and marble pick up was performed at the end of the session for ten repetitions.
  Interventions: Other: Resistance Exercises without Plyometric exercises

INTERVENTIONS:
Other: Resistance Exercises with Plyometric exercises — We will apply protocol for 8 weeks 24 Sessions (3 sessions in a week) and 10 sec rest between each segment, 3 sets of 10 repetitions.
  Resistive training will start in the form of manual resistive exercise for dorsiflexion, plantar flexion, eversion and inversion (manual resistance was applied for 3 to 5 seconds for ten repetitions in each cardinal plane).After resistance training the athletes will go for plyometric exercises and will follow the following guidelines.Tubing Exercises,Plyometric Ankle Jumps Ankle Circles
  Arms: Resistance Exercises with Plyometric exercises
Other: Resistance Exercises without Plyometric exercises — We will apply protocol for 8 weeks 24 Sessions (3 sessions in a week) and 10 sec rest between each segment, 3 sets of 10 repetitions. Resistive training will start in the form of manual resistive exercise for dorsiflexion, plantar flexion, eversion and inversion (manual resistance was applied for 3 to 5 seconds for ten repetitions in each cardinal plane). While controlling the time that a maximal contraction will be maintained, the therapist will assure that the targeted musculature will being maximally loaded
  Arms: Resistance Exercises without Plyometric exercises

SUMMARY:
Chronic ankle instability is characterized by a patient's being more than 12 months removed from the initial LAS and exhibiting a propensity for recurrent ankle sprains, frequent episodes or perceptions of the ankle giving way, and persistent symptoms such as pain, swelling, limited motion, weakness, and diminished self-reported function. This study will Compare Resistance Training with and without Plyometric exercises on Athletes with Chronic Ankle instability and changes will be recorded using different methods and tools. Patients will be randomly allocated into two different groups. Group A will be treated with resistance training and Group B will be treated with resistance training along with plyometric exercises . Participants will complete clinician-oriented tests. Participants of both groups will be evaluated before and after the application of respective interventions at the end of 8th week. Data will be analysed.

DETAILED DESCRIPTION:
Resistance training applies effort to overcome resistance, which results in increased muscle fibre recruitment and stronger synchronization, ultimately enhancing neuromuscular control and leading to muscular growth. Elastic resistance training is not only the cheaper intervention but is also able to promote similar strength gains to conventional resistance training. Both isokinetic muscle strength training and Thera-Band strength training have been used extensively to increase muscle strength after sports injuries and improve muscle performance in athletes, thereby accelerating injury recovery. Plyometric training provided benefits in both static and dynamic balances for individuals with Functional ankle instability. Plyometric are more effective than resistive exercises in improving functional performance of athletes after lateral ankle sprain. Convenient sampling technique will be used to collect the data. The sample size of 24 patients will be recruited. Patients will be randomly allocated into two different groups through sealed envelope method.12 patients will be allocated in each group A will be treated with resistance training and Group B will be treated with resistance training along with plyometric exercises so resistance training exercises are help full in athletic performance .Group B will be treated with resistance training along with plyometric exercises . Participants will complete patient-oriented questionnaires (CAIT for measuring the severity of functional ankle instability Foot and Ankle Ability Measure [FAAM] to assess physical function for individuals with foot and ankle related impairments, Numeric pain rating scale for pain, Short-Form 36 [SF-36] to indicate the health status of particular populations, to help with service planning and to measure the impact of clinical and social interventions. Culture-specific data are required to calculate SF-36 norm-based. Goniometer to measure available ranges will also be used Participants of both groups will be evaluated before the application of interventional techniques and re-evaluated after the application of respective interventions at the end of 8th week. Data will be analysed on SPSS 21 .The combination of both resistance and plyometric exercises could give more significant result.

ELIGIBILITY:
Inclusion Criteria:

* A history of at least 1 substantial ankle sprain with associated inflammatory symptoms and at least 1 interrupted day of desired physical activity, multiple episodes of the ankle "giving way," recurrent sprain, and "feelings of instability" in the 6 months before the study. Patients scoring the FAAM, there should be two scores, less than the ADL subscale and the Sports subscale, 20/21 items and 7/8 items must be completed, respectively
* If both ankles qualified, the ankle with the highest score (i.e. the most severely affected ankle) was considered the involved limb.

Exclusion Criteria:

* Volunteers were excluded if they had sustained an acute lower extremity injury in the 3 months before the study
* Having participated in formal rehabilitation in the 3 months before the study
* Having a history of lower extremity surgery or fracture that required alignment in the involved limb
* Having any diagnosed neurologic dysfunction, such as multiple sclerosis, Parkinson disease, or head injury.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 8 Weeks
  NPRS consists of a scale with 0-10 readings. The zero denotes no pain while 1, 2, 3 denotes to mild pain, 4, 5, 6 denotes to moderate pain while 7-10 denotes to severe pain.
Goniometer | 8 Weeks
  Active Range of Motion of the patient will be assessed using universal standard goniometer for ankle plantar flexion, dorsiflexion, inversion and eversion. All ranges will be assessed in sitting position.The data will be collected at baseline ankle goniometry. Goniometry will be performed using a universal goniometer with a measuring scale marked out at two-degree interval
The Star Excursion Balance Test (SEBT) | 8 Weeks
  The Star Excursion Balance Test (SEBT) is a widely accepted method of assessing dynamic postural stability. The Y Balance Test (YBT) is a commercially available device for measuring balance that uses 3 (anterior, posteromedial, and posterolateral) of the 8 SEBT directions and has been advocated as a method for assessing dynamic balance.
1 RM Leg Press test | 8 Weeks
  A training load that corresponds to 60-80% of one repetition maximum to increase muscle strength in leg and ankle of subjects with a loading range of 10-12 repetitions. It will measure the strength in pre treatment and post treatment evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Atif Javed, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex, Pakistan sports board complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanen L, Docherty CL, Van Der Pol B, Simon J, Schrader J. Prevalence of chronic ankle instability in high school and division I athletes. Foot Ankle Spec. 2014 Feb;7(1):37-44. doi: 10.1177/1938640013509670. Epub 2013 Nov 27. PMID 24287210
- [Background] Brown CN, Mynark R. Balance deficits in recreational athletes with chronic ankle instability. J Athl Train. 2007 Jul-Sep;42(3):367-73. PMID 18059992
- [Background] Chan KW, Ding BC, Mroczek KJ. Acute and chronic lateral ankle instability in the athlete. Bull NYU Hosp Jt Dis. 2011;69(1):17-26. PMID 21332435
- [Background] Yu P, Mei Q, Xiang L, Fernandez J, Gu Y. Differences in the locomotion biomechanics and dynamic postural control between individuals with chronic ankle instability and copers: a systematic review. Sports Biomech. 2022 Apr;21(4):531-549. doi: 10.1080/14763141.2021.1954237. Epub 2021 Aug 19. PMID 34412557
- [Background] Hall EA, Docherty CL, Simon J, Kingma JJ, Klossner JC. Strength-training protocols to improve deficits in participants with chronic ankle instability: a randomized controlled trial. J Athl Train. 2015 Jan;50(1):36-44. doi: 10.4085/1062-6050-49.3.71. Epub 2014 Nov 3. PMID 25365134
- [Background] Anderson K, Behm DG. The impact of instability resistance training on balance and stability. Sports Med. 2005;35(1):43-53. doi: 10.2165/00007256-200535010-00004. PMID 15651912
- [Background] Fakontis C, Iakovidis P, Kasimis K, Lytras D, Koutras G, Fetlis A, Algiounidis I. Efficacy of resistance training with elastic bands compared to proprioceptive training on balance and self-report measures in patients with chronic ankle instability: A systematic review and meta-analysis. Phys Ther Sport. 2023 Nov;64:74-84. doi: 10.1016/j.ptsp.2023.09.009. Epub 2023 Sep 30. PMID 37801793
- [Background] Wang B, Zhang X, Zhu F, Zhu W, Wang X, Jia F, Chen W, Zhang M. A randomized controlled trial comparing rehabilitation with isokinetic exercises and Thera-Band strength training in patients with functional ankle instability. PLoS One. 2022 Dec 1;17(12):e0278284. doi: 10.1371/journal.pone.0278284. eCollection 2022. PMID 36454876
- [Background] Lee HM, Oh S, Kwon JW. Effect of Plyometric versus Ankle Stability Exercises on Lower Limb Biomechanics in Taekwondo Demonstration Athletes with Functional Ankle Instability. Int J Environ Res Public Health. 2020 May 22;17(10):3665. doi: 10.3390/ijerph17103665. PMID 32456048
- [Background] Ismail MM, Ibrahim MM, Youssef EF, El Shorbagy KM. Plyometric training versus resistive exercises after acute lateral ankle sprain. Foot Ankle Int. 2010 Jun;31(6):523-30. doi: 10.3113/FAI.2010.0523. PMID 20557819
- [Background] Luan L, Adams R, Witchalls J, Ganderton C, Han J. Does Strength Training for Chronic Ankle Instability Improve Balance and Patient-Reported Outcomes and by Clinically Detectable Amounts? A Systematic Review and Meta-Analysis. Phys Ther. 2021 Jul 1;101(7):pzab046. doi: 10.1093/ptj/pzab046. PMID 33517464
- [Background] Molla-Casanova S, Ingles M, Serra-Ano P. Effects of balance training on functionality, ankle instability, and dynamic balance outcomes in people with chronic ankle instability: Systematic review and meta-analysis. Clin Rehabil. 2021 Dec;35(12):1694-1709. doi: 10.1177/02692155211022009. Epub 2021 May 31. PMID 34058832
- [Background] Matheny LM, Clanton TO. Rasch Analysis of Reliability and Validity of Scores From the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2020 Feb;41(2):229-236. doi: 10.1177/1071100719884554. Epub 2019 Oct 30. PMID 31665926
- [Background] Lins-Kusterer L, Valdelamar J, Aguiar CVN, Menezes MS, Netto EM, Brites C. Validity and reliability of the 36-Item Short Form Health Survey questionnaire version 2 among people living with HIV in Brazil. Braz J Infect Dis. 2019 Sep-Oct;23(5):313-321. doi: 10.1016/j.bjid.2019.08.001. Epub 2019 Sep 3. PMID 31491370